CLINICAL TRIAL: NCT07263542
Title: Effects of Body Weight Supported Treadmill Training on Motor Development in Patients Withh Dyskinetic Cerebral Palsy
Brief Title: Effects of Body Weight Supported Treadmill Training on Motor Development in Patients With Dyskinetic Cerebral Palsy
Acronym: BWSTT DCP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Principal Investigator, Prof. Dr. Shoaib Waqas, research supervisor, Lahore University of Biological and Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UBS24LMSPT011
Record Dates: First submitted 2025-11-16; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Cerebral Palsy (CP)
Keywords: cerebral palsy, BWSTT, DCP, RCT
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: The study utilizes parallel study design in which two groups will receive two different interventions. This design allows the comparison of two different treatment approaches under identical conditions.2
Who Masked: Outcomes Assessor
Masking Description: It will be a single-blinded RCT in which the outcome assessor will be kept blind about participants' allocation group. Assessor will be kept isolated from the intervention administration team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BWSTT (Experimental): Experimental group will recieve body weight supported treadmill training.
  Interventions: Other: BODY WEIGHT SUPPORTED TREADMILL TRAINING
- BOBATH (Active Comparator): comparator group will recieve Bobath therapy
  Interventions: Other: BOBATH THERAPY

INTERVENTIONS:
Other: BODY WEIGHT SUPPORTED TREADMILL TRAINING — The experimental group, will receive BWSTT with 40% weight offloading and a treadmill speed of 0.4 miles per hour (mph) at the start of the treatment. Weight offloading will be progressively decreased by 10% each week, leading to 30% offloading in the 2nd week, with the treadmill speed adjusting to 0.8 mph, 20% offloading in the 3rd week, with speed increasing to 1.2 mph; and 10% offloading during the 4th week of the intervention at a speed of 1.6 mph, for 30 minutes a day, five days a week for four weeks.
  Arms: BWSTT
Other: BOBATH THERAPY — The control group, will receive Bobath Therapy. The protocol will include dynamic balance training on a balance board for 6 minutes, followed by a 2-minute rest. Functional reaching and ball-throwing exercises for 6 minutes, followed by a 2-minute rest period. Supine pelvic bridging exercises for 6 minutes, followed by 2-minute rest intervals. weight-bearing exercises in sitting, standing, kneeling, and crawling positions to facilitate equal body weight transfers without disturbing postural control for another six minutes, followed by a 2-minute rest. Obstacle negotiation (cones, steps) with focus on: Heel-strike initiation, Stance-phase knee control, and Push-off symmetry for six minutes.
  Arms: BOBATH

SUMMARY:
This randomized controlled trial will evaluate motor development outcomes in children aged 5-12 years with dyskinetic cerebral palsy. The Primary Outcome measures will be Gross motor development, gait, trunk control, balance, and coordination, and will be assessed using the Shoaib Sensorimotor Development Tool (SMDT), Gross Motor Function Measure-88 (GMFM-88), Jacks' observational Gait Analysis scale, Trunk Impairment Scale (TIS), Time Up and Go Test, and Heel-to-Shin test. The fine motor development as a secondary outcome measure will be assessed using the Box and Block Test (BBT). Before allocating participants within the study, informed consent will be obtained to ensure rigorous adherence to the Principles of Ethical Research as outlined in the Helsinki Declaration for Ethical Research. Baseline readings will be recorded using the selected tools against the pre-defined outcome measures. Randomization will be done through an online tool, and the Participants will be divided into two intervention arms. The control group will receive conventional Bobath therapy, and the experimental group will undergo body weight-supported treadmill training (BWSTT), with both interventions administered over a period of 4 weeks, 5 days a week. Each session will be structured as follows: 5 minutes of warm-up exercises to prepare the body, followed by a 30-minute core treatment session focused on therapeutic interventions, concluding with 5 minutes of cooldown exercises to promote recovery and relaxation. This sequence ensures a balanced approach while maintaining the total session duration of 40 minutes, 5 days a week for 4 weeks. Statistical analysis of the results will be conducted using SPSS software to determine the significance of the findings. The Shapiro-Wilk test will be employed to determine the normality of the data. If the data distribution is normal, an independent t-test will be employed for between-group comparison; otherwise, non-parametric alternatives will be applied. Within group analysis, a paired t-test will be applied to evaluate differences and the results will be reported.

DETAILED DESCRIPTION:
The interventions to both groups will be applied for 40 minutes, 5 days a week, for 4 weeks. 5 minutes of warm-up and cool-down exercises will be administered to both groups before and after the administration of interventions. Subsequently, participants will receive 30 minutes of treatment according to the pre-designed protocol.

* Group A, or the experimental group, will receive BWSTT with 40% weight offloading and a treadmill speed of 0.4 miles per hour (mph) at the start of the treatment.
* Weight offloading will be progressively decreased by 10% each week, leading to 30% offloading in the 2nd week, with the treadmill speed adjusting to 0.8 mph
* 20% offloading in the 3rd week, with speed increasing to 1.2 mph; and 10% offloading during the 4th week of the intervention at a speed of 1.6 mph, for 30 minutes a day, five days a week for four weeks.

  40-minute BWSTT treatment sessions will have 8 minutes of exercise intervals followed by 2-minute rest intervals (16).

In contrast, GROUP-B or the control group will be given Bobath therapy.

* This will include dynamic balance training on a balance board for 6 minutes, followed by a 2-minute rest.
* functional reaching, and ball-throwing exercises for 6 minutes, followed by a 2-minute rest period.
* Supine pelvic bridging exercises for 6 minutes, followed by a 2-minute rest interval.
* weight-bearing exercises in sitting, standing, kneeling, and crawling positions to facilitate equal body weight transfers without disturbing postural control for another six minutes, followed by two minutes of rest.
* Obstacle negotiation (cones, steps) with focus on: Heel-strike initiation, Stance-phase knee control, and Push-off symmetry for six minutes.

ELIGIBILITY:
Inclusion Criteria:

- This study will include DCP Patients aged 5-12 years without any gender preference, falling at GMFCS levels I-II. The included participants must be capable of following instructions and must not have any known surgical or medical history.

Exclusion Criteria:

* DCP patients having cardiac complications, Past surgical history, Mental retardation, visual and cognitive deficits, under another gait training protocol, Congenital musculoskeletal defects, dislocations of the hip, significant hip and knee contractures, Behavioral disorders, or a history of Recent botulinum toxin injections, or uncontrolled epilepsy will be excluded from the study.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Gross motor Development | 4 weeks
  Gross Motor Development will be analyzed using GMFM-88. The tool categorizes motor development into five domains: lying and rolling, sitting, crawling and kneeling, standing, and walking, running, and jumping. These domains encompass 88 items, each scored on a 4-point ordinal scale ranging from 0 (indicating the inability to initiate the movement) to 3 (representing task completion). Higher scores reflect greater motor development in the patient.
Gross motor Development | 4 weeks
  Gross Motor Development will be analyzed using the Shoaib sensorimotor Development Tool. The standardized protocol comprises 72 developmentally stratified items employing a tripartite scoring matrix (0, 0.5, 1). The maximum attainable score is 72, while a score below 36 predicts atypical development.
Gait analysis | 4 week
  Gait analysis will be conducted using Jacks' Observational Gait Analysis. It is a qualitative assessment instrument designed for the systematic identification of pathokinematic deviations from normal gait patterns across the entire cycle. Instead of employing an ordinal quantification system, it employs a comparative observational framework where abnormalities are evaluated against established normative biomechanical parameters.
trunk control | 4 weeks
  Trunk Control assessment will be done using Trunk Impairment Scale. It assesses trunk control in three key domains: static sitting balance (ability to maintain upright posture), dynamic sitting balance (weight-shifting and reaching), and coordination (rotational movements). Scoring ranges from 0 (severe impairment) to 23 (normal function), providing quantitative data for rehabilitation progress tracking
Dynamic Balance and functional mobility | 4 weeks
  The balance will be assessed using Time up and Go Test. Key metrics measured are the time taken to stand, walk, turn, and sit. Normal score falls between 10-12 seconds. The greater the time required to accomplish the task, the greater the gravity of the problem.
motor coordination assessment | 4 weeks
  Motor coordination assessment will be conducted through the standardized heel-shin coordination test to evaluate volitional limb control precision. Participants will be instructed to perform the maneuver in supine position by sliding the plantar aspect of one foot along the contralateral tibial crest, maintaining continuous contact from the tibial tuberosity to the lateral malleolus. The quality of the movement will be indicative of coordinated limb function. Jerky or clumsy movement and failure to perform it throughout the dictated range are indicative of neurological pathology.

SECONDARY OUTCOMES:
Fine Motor Development | 4 weeks
  Fine Motor Development will be assessed through the Box and Block Test by counting the number of small blocks a person can move from one side of a partitioned box to the other in 60 seconds. A higher score indicates greater dexterity, while a lower score may suggest impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Hafsa Jamil, DPT, Principal Investigator — Lahore University of Biological and Applied Sciences
Locations (1):
- University of Biological and Applied Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual patient data (IDP) will not be disclosed to preserve patient confidentiality and comply with privacy protection protocols. Sharing raw datasets carries inherent risks, including potential misinterpretation of sensitive health information and unauthorized utilization by third parties, which could lead to non-consensual exploitation or breaches of ethical guidelines. To mitigate these concerns, aggregated or anonymized data will be provided in alignment with regulatory standards for transparency while safeguarding participant identities.